CLINICAL TRIAL: NCT05088902
Title: Pilot Testing Manual For Validation Purposes Providing Clearance for COVID-19 Tested Individuals Using the TERA Bio Station T101
Brief Title: Validation of TERA Bio Station T101 of COVID-19 Tested Population.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tera Group (Industry)
Responsible Party: Sponsor
Other Study IDs: Validation of TERA Bio Station
Record Dates: First submitted 2021-10-21; First posted 2021-10-22 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: TERABio Ltd. — Covid- 19 investigational breath test compared to RT- PCR test. TERABio Ltd. has developed a rapid screening tool intended to determine if a tested individual is COVID-19-free (Negative to COVID-19 ).

SUMMARY:
TERABio Ltd. has developed a rapid screening tool intended to determine if a tested individual is COVID-19-free (Negative to COVID-19).

DETAILED DESCRIPTION:
The goal of the pilot is to perform a localized validation to the TERA Bio Tests by TERA Bio Station(s). Success Criteria: Clearing at least 80% of the healthy population.

Pilot duration: approx. 6-10 work weeks long.

Research Population Requirements:

Male and Female, age ≥ 18 years old, whose COVID-19 virus infection status is known and verified for at least the last 24 hours (prior to the TERA.Bio test).

The study will include a minimum of 300 tested Positive individuals and a minimum of 700 Negative individuals, tested during the 24 hours prior to the TERA.Bio test.

Additional PCR tests on specific individuals, based on their symptomatic status and/or their PCR's CT value may be required be done 3 days after taking the breath test.

It is expected that each day will contain both Positive and Negative individuals in a similar ratio to the overall expected one (30%).

Test Procedure:

A staff member will explain to the tested individual about the test and will hand him an informed consent form. The tested individual will review and sign the consent form and return it to the staff member. The individual must sign the informed consent form in order to participate in the pilot testing. The individual's breath sample is then taken by blowing three times into a disposable TERATube. Thereafter, the tube is sealed, sterilized, and scanned by the TERA Bio Station for analysis of its bio-chemical spectral signature.

Blind Test objectives and method:

Following data analytics of the previous phase and once achieving sufficient testing, a blind test may be performed to validate the accuracy of the TERA.Bio test. The blind test will include 60 individuals from which 30 must be Positive for COVID-19.

The blind test's tested individuals will be tested in the exact way the pilot testing was performed and with RT-PCR with the exact same CT.

TERA.Bio's team will conduct the breath tests scanning and decoding procedure without obtaining the RT-PCR results in-advance.

The TERA.Bio team will send predictions for each tested individual (suspected\negative) to the pilot manager and primary investigator after ALL pilot participants have been tested.

The RT-PCR results will then be sent to the TERA.Bio team. The two parties will compare the results obtained from the TERA Bio Station to the results from the RT-PCR.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old (under 18 years old - only if it is allowed under local regulations and with legal guardian's approval and consent if needed.
2. COVID-19 virus infection status is known and verified 24 hours prior to a TERA.Bio test by RT-PCR and if required, a repeated PCR test based on symptomatic status and or / the CT value of the tested individual.
3. Signed Informed consent form.

Exclusion Criteria:

1. Discrepancies to inclusion criteria
2. Individuals under general anaesthesia
3. Individuals lacking the capability to personally sign the consent form.
4. Individuals lacking the capability to exhale breath.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Research Population Requirements:
  * Male and Female, age ≥ 18 years old, whose COVID-19 virus infection status is known and verified for at least the last 24 hours (prior to the TERA.Bio test).
  * The study will include a minimum of 300 tested Positive individuals and a minimum of 700 Negative individuals, tested during the 24 hours prior to the TERA.Bio test.
  * Additional PCR tests on specific individuals, based on their symptomatic status and/or their PCR's CT value may be required be done 3 days after taking the breath test.
  * It is expected that each day will contain both Positive and Negative individuals in a similar ratio to the overall expected one (30%)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-03-06 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Clearing at least 80% of the healthy population | 7 Weeks (Estimated)
  TERABio Ltd. has developed a rapid screening tool intended to determine if a tested individual is COVID-19-free (Negative to COVID-19).
  The goal of the pilot is to perform a localized validation to the TERA Bio Tests by TERA Bio Station(s)- Success Criteria -Clearing at least 80% of the healthy population.

CONTACTS AND LOCATIONS:
Overall Officials: Nihat Müjdat Hökenek, MD, Principal Investigator — TR Ministry of Health Istanbul Provincial Health Directorate Kartal Dr. Lütfi Kirdar City Hospital
Locations (1):
- TR Ministry of Health Istanbul Provincial Health Directorate Kartal Dr. Lütfi Kirdar City Hospital, Istanbul, Turkey (Türkiye)